CLINICAL TRIAL: NCT06642766
Title: Open Label Study of a Novel, Commercially Available Fiber Product for Gas, Bloating, and Bowel Regularity
Brief Title: Fiber Product for Gas, Bloating, and Bowel Regularity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bell Cinical Service (Industry)
Collaborators: LX Medical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20243173
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Bloating; Bowel Irregularities; Bowel Gas
Keywords: fiber supplement; bloating; nutralieve; Microbiome; Gut microbiota; irregular bowel movements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fiber supplemenmt (Experimental)
  Interventions: Dietary Supplement: Fiber supplement

INTERVENTIONS:
Dietary Supplement: Fiber supplement — Subjects that meet the inclusion criteria and with symptoms appropriate for fiber supplementation are eligible to participate. Participants will be instructed to use the fiber product (NutraLieve) as currently labeled; start with a dosage of 4-5 grams per day (one heaping teaspoon), initially taken once daily, increasing up to 3 heaping teaspoons a day (maximum dose 15 grams/day) on an as needed basis.Participants will be prospectively assessed for symptoms at baseline and at 6 weeks.
  * The primary endpoint, number of bowel movements, will be assessed by bowel movements in the last 72-hour period at baseline and at 6 weeks, by patient recall/diary.
  * Secondary endpoints, reduction in bloating or gas, or any adverse events will be assessed using analog scales, also by 72-hour recall at baseline and at 6 weeks, by patient recall/diary.

SUMMARY:
This is a new, commercially available, over-the-counter fiber supplement that combines 8 fibers. The varied nature of the fibers in this product is designed to create a more diverse microbiome (bacteria that live within the human GI tract). In general, the more diverse the microbiome the less inflammatory the gut. The purpose of this study is to evaluate the effects of a new fiber product on bloating, gas, and bowel movements.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have experienced two or more of the following criteria for at least 3 months with symptom onset at least 6 months prior: straining during at least 25% of defecations, lumpy or hard stools in at least 25% of defecations, sensation of incomplete evacuation for at least 25% of defecations, sensation of anorectal obstruction/blockage for at least 25% of defecations, manual maneuvers to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvic floor), loose stools are rarely present without the use of laxatives Or,
* Subjects have experienced 2 or more of the following criteria of recurrent abdominal pain, for at least 3 months, with symptom onset at least 6 months prior: pain related to defecation, associated with a change in frequency of stool, associated with a change in form (appearance) of stool Or,
* Subjects have experienced 2 or more of the following criteria for at least 3 months, with symptom onset at least 6 months prior: recurrent abdominal pain, on average, at least 1 day per week in the last 3 months associated with two of the following criteria: pain related to defecation, pain associated with a change in frequency of stool and pain associated with a change in form (appearance) of stool.
* The subject predominantly experiences loose or watery stools (Bristol Stool Form Scale types 6-7), more than 25% of the time, or hard or lumpy stools (types 1-2) less than 25% of the time.
* The symptoms should be chronic and interfere with daily activities, cause worry or affect the quality of life.

Exclusion Criteria:

* Loose stools are present for more than 25% of defecations
* Unable to provide informed consent
* Hematochezia
* Prior colon surgery
* Thyroid disease
* Pelvic floor disorder
* Known allergies or intolerance to fiber products
* infectious diarrhea or food poisoning
* inflammatory bowel disease, including microscopic colitis
* fecal incontinence or rectal prolapse

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Number of bowel movement | 6 weeks
  - The primary endpoint, number of bowel movements, will be assessed by bowel movements in the last 72-hour period at baseline and at 6 weeks, by patient recall/diary.

SECONDARY OUTCOMES:
Bloating | 6 weeks
  - Reduction in bloating will be assessed using analog scales, also by 72-hour recall at baseline and at 6 weeks, by patient recall/diary.
Gas | 6 weeks
  Reduction in gas will be assessed using analog scales, also by 72-hour recall at baseline and at 6 weeks, by patient recall/diary.

CONTACTS AND LOCATIONS:
Locations (1):
- XL Medical, Edina, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Subject's demographics and measured outcomes
Supporting Information: Study Protocol